CLINICAL TRIAL: NCT02137733
Title: The Cardiac Insufficiency BIsoprolol Study in Japanese Patients With Chronic Heart Failure (CIBIS-J)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mebix Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ji 012-0386
Record Dates: First submitted 2014-05-01; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Bisoprolol; Carvedilol

ARMS (2):
- Bisoprolol group (Active Comparator): Daily oral administration of bisoprolol 0.625 mg tablet once a day should be given (Step 1). If tolerability is confirmed by an investigator, the dose should be increased to 1.25 mg (bisoprolol 0.625 mg, 2 tablets; or bisoprolol 2.5 mg, half tablet; once daily) (Step 2). In the same manner, the doses should be increased to 2.5 mg (bisoprolol 2.5 mg, 1 tablet; or bisoprolol 5 mg, half tablet; once daily, Step 3), to 3.75 mg (bisoprolol 2.5 mg, 1.5 tablets once daily, Step 4), and to 5 mg (bisoprolol 2.5 mg, 2 tablets; or bisoprolol 5 mg, 1 tablet; once daily, Step 5).
  Interventions: Drug: Bisoprolol
- Carvedilol group (Active Comparator): Daily oral administration of carvedilol 1.25 mg, 1 tablet twice a day (after breakfast and supper) should be given (Step 1). If tolerability is confirmed by an investigator after administering 2.5 mg/day of carvedilol, the dose should be increased to 5 mg (carvedilol 2.5 mg, 1 tablet twice daily) (Step 2). In the same manner, the dose should be increased to 10 mg (carvedilol 2.5 mg, 2 tablets twice daily, Step 3), to 15 mg (carvedilol 2.5 mg, 3 tablets twice daily, Step 4), and to 20 mg (carvedilol 10 mg, 1 tablet twice daily, Step 5).
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Bisoprolol
  Arms: Bisoprolol group
Drug: Carvedilol
  Arms: Carvedilol group

SUMMARY:
The purpose of this study is to investigate the non-inferiority of bisoprolol to carvedilol by evaluating tolerability (The probability that administered maintenance dose reaches the maximum will be determined as an indicator) as a primary endpoint when bisoprolol or carvedilol is administered for 48 weeks to Japanese chronic heart failure patients. In addition, the safety and efficacy of bisoprolol will be investigated.

ELIGIBILITY:
Inclusion Criteria:

As a result of diagnosis and tests before registration, a patient who is considered by an investigator to meet all requirements and to have ability to consent can be enrolled.

1. Primary disease: In principle, ischemic heart disease or dilated cardiomyopathy.
2. Heart failure patients with 40% or less of left ventricular ejection fraction (LVEF) .
3. Patients in NYHA functional classification Class II, III, or IV (including a medical history).
4. Basic treatment: In principle, patients undergoing treatment with an ACE inhibitor (or angiotensin receptor blocker (ARB)), a diuretic, a digitalis preparation, etc.
5. Patients who had not undergone treatment with a beta-blocker (except eye drops) within 8 weeks before the registration date.
6. Age: Patients aged 20 to less than 85 on the day of obtaining written informed consent.
7. Hospitalized/outpatient: Either hospitalized or outpatient status.
8. Gender: Male or Female

Exclusion Criteria:

Patients who meet any of the following exclusion criteria at the time of registration will be excluded:

1. Patients who are considered not to be candidates for administration of bisoprolol or carvedilol.
2. Patients who have developed acute myocardial infarction within 8 weeks before the registration day.
3. Patients who have history of stroke or serious cerebrovascular accident within 1 year before the registration day.
4. Patients with poor prognosis and life-threatening disease, such as malignant tumor, or such medical history within 5 years before the registration day.
5. Patients who are scheduled to undergo coronary revascularization (Coronary artery bypass grafting; CABG, Percutaneous coronary intervention; PCI) during the study period.
6. Patients who are pregnant, lactating, may become pregnant, or want to become pregnant during the study.
7. Patients from whom written informed consent cannot be obtained.
8. Patients who are judged by an investigator to be inappropriate for this study for any other reason.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Tolerability: The probability that administered maintenance dose reaches the maximum (bisoprolol 5 mg/day, carvedilol 20 mg/day) | 48 weeks

SECONDARY OUTCOMES:
Efficacy: New York Heart Association (NYHA) Functional Classification | 24 and 48 weeks
Efficacy: Left Ventricular Ejection Fraction (LVEF) | 24 and 48 weeks
Efficacy: Left Ventricular End Diastolic Volume (LVEDV), Left Ventricular End Systolic Volume (LVESV) | 24 and 48 weeks
Efficacy: Heart rate | 24 and 48 weeks
Efficacy: Plasma brain natriuretic peptide (BNP) | 24 and 48 weeks
Safety: All deaths | 48 weeks
Safety: Deaths with cardiovascular causes | 48 weeks
Safety: Hospitalization for cardiovascular causes | 48 weeks
Safety: Exacerbation of heart failure, resulting in hospitalization, and/or intensification of treatment (increase in dose of any diuretics, vasodilators or cardiotonics, in comparison with the dose-setting period), or administration of new drugs. | 48 weeks
Safety: Deaths due to heart failure (pump-failure deaths, and deaths associated with exacerbation of heart failure) | 48 weeks
Safety: Sudden deaths, including deaths due to arrhythmia | 48 weeks
Safety: Deaths with non-cardiovascular causes | 48 weeks
Safety: Adverse events | 48 weeks
Safety: Changes in clinical laboratory test results | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Tsutsui, Study Chair — Hokkaido University Graduate School of Medicine
Locations (110):
- Japan (110):
  - Banbuntane Hotokukai Hospital, Nagoya, Aichi-ken
  - Chukyo Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Takezawa Clinic, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Hirosaki University School of Medicine & Hospital, Hirosaki, Aomori
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Hakujyuji Hospital, Fukuoka, Fukuoka
  - Haradoi Hospital, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Chiyo Clinic, Kitakyushu, Fukuoka
  - Kitakyushu Municipal Yahata Hospital, Kitakyushu, Fukuoka
  - Takagi Hospital, Ōkawa, Fukuoka
  - Fukushima Daiichi Hospital, Fukushima, Fukushima
  - Ohara General Hospital, Fukushima, Fukushima
  - Gifu University Hospital, Gifu, Gifu
  - Kizawa memorial hospital, Minokamo, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi, Gunma
  - Maebashi Red Cross Hospital, Maebashi, Gunma
  - Ota Memorial Hospital, Fukuyama, Hiroshima
  - Hiroshima General Hospital of West Japan Railway Company, Hiroshima, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Shobara Red Cross Hospital, Shōbara, Hiroshima
  - Hokkaido P.W.F.A.C Asahikawa-Kosei General Hospital, Asahikawa, Hokkaido
  - Kihara cardiovascular clinic, Asahikawa, Hokkaido
  - Ebetsu City Hospital, Ebetsu, Hokkaido
  - Hokkaido Chuo Rosai Hospital, Iwami, Hokkaido
  - Otaru Kyokai Hospital, Otaru, Hokkaido
  - Hokkaido Medical Center, Sapporo, Hokkaido
  - JR Sapporo Hospital, Sapporo, Hokkaido
  - KKR Sapporo Medical Center, Sapporo, Hokkaido
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Sapporo Medical Center NTT East, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Sunagawa City Medical Center, Sunagawa, Hokkaido
  - Hyogo Brain and Heart Center, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Hyogo College Of Medicine, Nishinomiya, Hyōgo
  - Nishiwaki Municipal Hospital, Nishiwaki, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Kanazawa Cardiovascular Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University, Kita-gun, Kagawa-ken
  - Tenyoukai Central Hospital, Kagoshima, Kagoshima-ken
  - St. Marianna University School of Medicine, Kawasaki, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Nishi Yokohama Hospital, Yokohama, Kanagawa
  - Yokohamashintoshi Neurosurgical Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Takenaka Clinic, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki Goto Chuoh Hospital, Gotō, Nagasaki
  - Ebisu-hospital, Nagasaki, Nagasaki
  - Medical Inc. Kosei-kai Nijigaoka Hospital, Nagasaki, Nagasaki
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Nara Hospital Kinki University Faculty of Medicine, Ikoma, Nara
  - Nara Prefecture Western Medical Center, Ikoma, Nara
  - Nara Medical University, Kashihara, Nara
  - Nara City Hospital, Nara, Nara
  - Nara Prefecture General Medical Center, Nara, Nara
  - Tsunan Metropolitan Hospital, Nakauonuma-gun, Niigata
  - Kuwana hospital, Niigata, Niigata
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Ohama Daiichi Hospital, Naha, Okinawa
  - Urasoe General Hospital, Urasoe, Okinawa
  - Osaka National Hospital, Chuo, Osaka
  - Nozaki Tokushukai Hospital, Daitō, Osaka
  - Kansai Medical University Hirakata Hospital, Hirakata, Osaka
  - Graduate School of Medicine and Faculty of Medicine, Osaka, Osaka
  - JCHO Osaka Hospital, Osaka, Osaka
  - Kitano Hospital, Osaka, Osaka
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Yayoigaoka Kage Hospital, Tosu, Saga-ken
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Ikebukuro Hospital, Kawagoe, Saitama
  - Saitama Medical Center Jichi Medical University, Saitama, Saitama
  - Kusatsu General Hospital, Kusatsu, Shiga
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo Shizuoka Hospital, Izunokuni, Shizuoka
  - Dokkyo Medical University, Shimotsuga-gun, Tochigi
  - Ohta Clinic, Anan, Tokushima
  - Tokushima University Hospital, Tokushima, Tokushima
  - Nishiarai Heart Center Hospital, Adachi-ku, Tokyo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Medical Hospital of Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Fuchū, Tokyo
  - Minamino Heart Clinic, Hachiōji, Tokyo
  - Hino Municipal Hospital, Hino, Tokyo
  - Tokyo Medical Center, Meguro-ku, Tokyo
  - 100, Setagaya-ku, Tokyo
  - Daisankitashinagawa hospital, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Yamaguchi Grand Medical Center, Hōfu, Yamaguchi
  - Shimonoseki City Hospital, Shimonoseki, Yamaguchi
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Kanoiwa General Hospital, Yamanashi, Yamanashi